CLINICAL TRIAL: NCT01463059
Title: A Randomized, Double-blind, Placebo Controlled, Dose Ranging Study to Evaluate the Efficacy and Safety of CDP6038 Administered Subcutaneously for 12 Weeks to Asian Subjects With Active Rheumatoid Arthritis Having Previously Failed TNF Blocker Therapy
Brief Title: Efficacy and Safety of Olokizumab With Rheumatoid Arthritis With Previously Failed to Anti-tumor Necrosis Factor (Anti-TNF) Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA0083
Record Dates: First submitted 2011-10-27; First posted 2011-11-01 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Monoclonal Antibody; Interleukin-6; Olokizumab; CDP6038
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — olokizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo every 2 weeks (Placebo Comparator): Injections administered at week 0, 2, 4, 6, 8 and 10
  Interventions: Biological: Placebo
- Olokizumab 60 mg every 2 weeks (Experimental): Olokizumab 60 mg injections administered at week 0, 2, 4, 6, 8 and 10
  Interventions: Biological: Olokizumab 60 mg
- Olokizumab 60 mg every 4 weeks (Experimental): Olokizumab 60 mg injection administered at week 0, 4, and 8 and Placebo injection administered at week 2, 6, and 10
  Interventions: Biological: Placebo; Biological: Olokizumab 60 mg
- Olokizumab 120 mg every 2 weeks (Experimental): Olokizumab 120 mg injections administered at week 0, 2, 4, 6, 8 and 10
  Interventions: Biological: Olokizumab 120 mg
- Olokizumab 120 mg every 4 weeks (Experimental): Olokizumab 120 mg injections administered at week 0, 4 and 8 and Placebo injections at week 2, 6 and 10
  Interventions: Biological: Placebo; Biological: Olokizumab 120 mg
- Olokizumab 240 mg very 4 weeks (Experimental): Olokizumab 240 mg injections administered at week 0, 4 and 8 and Placebo injections at week 2, 6 and 10
  Interventions: Biological: Placebo; Biological: Olokizumab 240 mg

INTERVENTIONS:
Biological: Placebo — Placebo solution for injection, administered as subcutaneous injections
  Arms: Olokizumab 120 mg every 4 weeks; Olokizumab 240 mg very 4 weeks; Olokizumab 60 mg every 4 weeks; Placebo every 2 weeks
Biological: Olokizumab 60 mg — Olokizumab 60 mg solution for injection, administered as subcutaneous injections
  Other Names: CDP6038
  Arms: Olokizumab 60 mg every 2 weeks; Olokizumab 60 mg every 4 weeks
Biological: Olokizumab 120 mg — Olokizumab 120 mg solution for injection, administered as subcutaneous injections
  Other Names: CDP6038
  Arms: Olokizumab 120 mg every 2 weeks; Olokizumab 120 mg every 4 weeks
Biological: Olokizumab 240 mg — Olokizumab 240 mg solution for injection, administered as subcutaneous injections
  Other Names: CDP6038
  Arms: Olokizumab 240 mg very 4 weeks

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of CDP6038 administered subcutaneous (sc) at various doses compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of adult-onset RA of at least 6 months' (24 weeks) duration as defined by the 1987 ACR classification criteria or a score of ≥6 as defined by the ACR/European League Against Rheumatism Classification and Diagnostic Criteria for RA
* Must have moderately to severely active RA disease as defined by ≥6 tender joints (68-joint count) at Screening and Baseline, ≥6 swollen joints (66-joint count) at Screening and Baseline, CRP ≥1.2 times the upper limit of normal (ULN) or ESR >28mm/hour
* Must be on an MTX dose of 6 to 16mg/week in Japan or 7.5 to 20mg/week in Korea and Taiwan, which has been stable for at least 6 weeks prior to Screening with a stable route of administration
* Must have had intolerance or inadequate response to treatment with 1 or more TNF-blocker therapies within 2 years of Screening
* Female subjects must be either postmenopausal for at least 1 year, surgically incapable of childbearing, or effectively practicing 2 acceptable methods of contraception

Exclusion Criteria:

* Have a diagnosis of any other inflammatory arthritis
* Female subjects who are breast-feeding, pregnant, or plan to become pregnant during the study or within 24 weeks
* Disease modifying antirheumatic drug (DMARDs) other than methotrexate (MTX)
* Subjects with known concurrent acute or chronic viral hepatitis B or C infection
* Subject has known tuberculosis (TB) disease, high risk of acquiring TB infection, or latent TB infection
* Subjects with known history of or current clinically active infection
* Subjects at high risk of infection
* Subjects with known human immunodeficiency virus (HIV) or human T cell lymphotropic virus type 1 (HTLV 1) infection
* Have received vaccinations within 8 weeks prior to Screening or plan to receive vaccines during the study (with the exception of injectable influenza and pneumococcal vaccinations which are permitted)
* Concurrent malignancy or a history of malignancy (with the exception of successfully treated carcinoma of the cervix more than 5 years prior to Screening or no more than 2 successfully treated basal cell carcinomas within 2 years prior to Screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Disease Activity Score 28-joint count (C-reactive protein) (DAS28[CRP]) at Week 12 | From Week 0 (Baseline) to Week 12

SECONDARY OUTCOMES:
Number of responders in American College of Rheumatology 20% Response Criteria (ACR20) at Week 12 | From Week 0 (Baseline) to Week 12
  Number of subjects who achieve ACR 20 will be calculated at week 12. The calculation is based on the improvement from the baseline in the number of tender joints and in the number of swollen joints each; and the improvement based on assessments from the patient and the physician drawn according to defined standards.
Number of responders in American College of Rheumatology 50% Response Criteria (ACR50) at Week 12 | From Week 0 (Baseline) to Week 12
  Number of subjects who achieve ACR 50 will be calculated at week 12. The calculation is based on the improvement from the baseline in the number of tender joints and in the number of swollen joints each; and the improvement based on assessments from the patient and the physician drawn according to defined standards.
Number of responders in American College of Rheumatology 70% Response Criteria (ACR70) at Week 12 | From Week 0 (Baseline) to Week 12
  Number of subjects who achieve ACR 70 will be calculated at week 12. The calculations is based on the improvement from the baseline in the number of tender joints and in the number of swollen joints each; and the improvement based on assessments from the patient and the physician drawn according to defined standards.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (39):
- Japan (23):
  - 102, Chiba
  - 114, Fukuoka
  - 115, Fukuoka
  - 113, Hiroshima
  - 120, Kakogawa
  - 118, Kumamoto
  - 116, Kurume
  - 121, Matsuyama
  - 122, Matsuyama
  - 107, Nagaoka
  - 110, Nagoya
  - 103, Narita
  - 112, Okayama
  - 119, Ōita
  - 100, Sapporo
  - 117, Sasebo
  - 124, Tokorozawa
  - 123, Tokyo
  - 101, Tomakomai
  - 108, Tonami
  - 111, Tsu
  - 105, Yokohama
  - 104, Yotukaido
- South Korea (5):
  - 200, Daejeon
  - 201, Junggu
  - 202, Seongdong-gu
  - 203, Seoul
  - 204, Seoul
- Taiwan (11):
  - 303, Changhua
  - 304, Dalin-Town
  - 305, Hualien City
  - 300, Kaohsiung City
  - 301, Taichung
  - 306, Taichung
  - 307, Taichung
  - 302, Taipei
  - 308, Taipei
  - 309, Taipei
  - 310, Taipei

REFERENCES:
- [Derived] Takeuchi T, Tanaka Y, Yamanaka H, Amano K, Nagamine R, Park W, Shiozawa K, Tsukano M, Wei JC, Shao J, Togo O, Mashimo H. Efficacy and safety of olokizumab in Asian patients with moderate-to-severe rheumatoid arthritis, previously exposed to anti-TNF therapy: Results from a randomized phase II trial. Mod Rheumatol. 2016;26(1):15-23. doi: 10.3109/14397595.2015.1074648. Epub 2015 Sep 10. PMID 26358841